CLINICAL TRIAL: NCT05731050
Title: A Phase II, Open Label, Multi Dose Study of NM8074 in Soliris-Treated Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Study of NM8074 in Soliris-Treated Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovelMed Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NM8074-PNH-101
Record Dates: First submitted 2023-02-01; First posted 2023-02-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: PNH - Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Intervention Model Description: A total of at least 6 patients (maximum of 10) with documented PNH and at least 3 months of Soliris treatment prior to Screening will be enrolled at the study site. The total duration of study term participation for all subjects will be up to 22 weeks, including a screening period of up to 8 weeks, a 12-week treatment period, and 2 weeks of a washout period. All subjects will receive a dose of 15 mg/kg NM8074 every two weeks with a total of 6 doses, from Day 1 to Day 84 during the treatment period. No more than two subjects will be dosed in a single day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NM8074 (Experimental): All subjects will receive a dose of 15 mg/kg NM8074 every two weeks with a total of 6 doses, from Day 1 to Day 84 during the treatment period.
  Interventions: Drug: NM8074

INTERVENTIONS:
Drug: NM8074 — NM8074 will be administered as an intravenous infusion. All enrolled subjects will receive a dose of 15 mg/kg NM8074 once every two weeks for a total of 6 doses from Day1 to Day 84.
  For Soliris-treated PNH subjects, admission and dosing of NM8074 on Day 1 should be scheduled to coincide with the next scheduled dose of Soliris (i.e., 14 ± 2 days after the last Soliris dose). Soliris should NOT be administered on Day 1 or at any time thereafter during course of the study.
  Subjects in the treatment groups will receive a dose of 15 mg/kg of NM8074 on Day 1, which will be administered during the study visit by the site staff. During the remainder of the treatment period, subjects will be given another 15 mg/kg dose every two weeks at approximately the same time. On days of scheduled study visits at the Investigation Site, the dose must be administered after blood work is completed.

SUMMARY:
The proposed study, NM8074-PNH-101, is a phase II, open-label, multi-dose, unicenter trial to evaluate the safety and efficacy of NM8074 in Soliris-treated PNH subjects.

DETAILED DESCRIPTION:
The proposed study, NM8074-PNH-101, will evaluate the safety and efficacy of NM8074 in Soliris-treated PNH subjects. The drug will be administered by intravenous (IV) infusion to adult patients who qualify based on the inclusion/exclusion criteria. A total of at least 6 patients (maximum of 10) with documented PNH and at least 3 months of Soliris treatment prior to Screening will be enrolled at the study site. The total duration of study term participation for all subjects will be up to 22 weeks, including a screening period of up to 8 weeks, a 12-week treatment period, and 2 weeks of a washout period. All subjects will receive a dose of 15 mg/kg NM8074 every two weeks with a total of 6 doses, from Day 1 to Day 84 during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years at the time of consent
* Confirmation of PNH diagnosis by flow cytometry evaluation of red blood cells (RBCs) and white blood cells (WBCs), with granulocyte or monocyte clone size of ~5%
* Presence of one or more of the following PNH-related signs or symptoms within 3 months of Screening: fatigue, hemoglobinuria, abdominal pain, shortness of breath (dyspnea), anemia: hemoglobin < 10 g/dL, history of a major adverse vascular event (including thrombosis), dysphagia, erectile dysfunction, PNH-mediated pRBC transfusions
* PNH patients must be undergoing treatment with Soliris for at least 3 months prior to screening, and must have a lactate dehydrogenase (LDH) level ≥ 1.5 times the upper limit of normal (ULN) during Screening
* Willing and able to understand and complete informed consent procedures, including signing and dating the informed consent form (ICF), and comply with the study visit schedule.
* Female subjects of childbearing potential must have a negative pregnancy test at Screening, and must not be planning pregnancy throughout the extent of the study term
* Female subjects of child-bearing potential and all male subjects must agree to use of effective contraception during study
* Soliris treated individuals must be able to provide documentation of vaccination against meningococcal infections.

Exclusion Criteria:

* Platelet count < 30,000/µL at Screening
* Absolute neutrophil count (ANC) < 500 cells/µL at Screening
* Body weight < 85 lbs. (38 kg) at Screening
* Estimated glomerular filtration rate of < 30 mL/min/1.73m2 based on modification of diet in renal disease (MDRD) equation, creatinine clearance, or CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) at Screening
* Elevation of liver function tests: alanine aminotransferase (ALT) > 2xULN or direct bilirubin and alkaline phosphatase (ALP) both > 2xULN
* Has a known history of meningococcal disease or N. meningitidis infection
* Has an immunological disorder, such as, but not limited to, human immunodeficiency virus (HIV) infection (as evident by HIV-1 or HIV-2 antibody titer) or any acute or chronic infection including, but not limited to, hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Currently active systemic infection or suspicion of active bacterial, viral, or fungal infection that requires antibiotic, antifungal, antiparasitic, or antiviral mediations
* Temperature > 38°C for more than two weeks prior to screening
* History of bone marrow or solid organ transplantation
* Pregnant, planning to become pregnant, or nursing female subjects
* Recent surgery requiring general anesthesia within the 2 weeks prior to Screening, or expected to have surgery requiring general anesthesia during the 12-week treatment period
* Active malignancy requiring surgery, chemotherapy, or radiation within the prior 12- months (subjects with a history of malignancy who have undergone curative resection or otherwise not requiring treatment for at least 12-months prior to screening with no detectable recurrences are allowed)
* History of any significant major medical conditions (cardiac, pulmonary, renal, e endocrine, or hepatic), or psychiatric disorder that, in the opinion of the Investigator, would make the subject unsuitable for participation in the study
* PNH patients currently under complement blocker treatments other than Soliris
* Concomitant use of anticoagulants is prohibited, if not on a stable regimen for at least 2 weeks prior to Day 1
* Participation in any experimental small molecule or non-antibody therapy within 60 days prior to dosing on Day 1 (participation in observational studies and/or registry studies is permitted)
* Known or suspected history of illegal recreational drug or alcohol abuse within 1 year prior to start of screening
* Hypersensitivity or history of allergy to excipients in NM8074 formulation
* Unable or unwilling to comply with the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Normalization of serum LDH(Lactate dehydrogenase) levels from baseline levels | Up to Week 12
Change from Baseline or Percent Change from Baseline in total hemoglobin levels (g/dL) | Up to Week 12
Change from Baseline or Percent Change from Baseline in total number of units of packed red blood cells (pRBCs) transfused through Week 12 | Up to Week 12
Change from Baseline or Percent Change from Baseline in number of transfusions | Up to Week 12
Percent Change from Baseline in Levels of Membrane Attack Complex (MAC) via Alternative Pathway (AP) of Complement Activity as Compared to Percent Change from Baseline in Levels of MAC via Classical Pathway (CP) of Complement Activity | Up to Week 12

SECONDARY OUTCOMES:
Normalization of anemia | Up to Week 12
  Change from Baseline or Percent Change from Baseline in Reticulocyte Count
Normalization of anemia | Up to Week 12
  Change from Baseline or Percent Change from Baseline in Bilirubin Levels
Change from Baseline or Percent Change from Baseline of C3b deposition on PNH Type II and Type III RBCs via Flow Cytometry | Up to Week 12

IPD SHARING:
Plan to Share IPD: No